CLINICAL TRIAL: NCT05020743
Title: A Natural History Study of Patients With Adult-Onset Leukoencephalopathy With Axonal Spheroids and Pigmented Glia (ALSP)
Brief Title: Natural History Study in Adult-Onset Leukoencephalopathy With Axonal Spheroids and Pigmented Glia
Acronym: ALSP
Status: Terminated | Type: Observational
Why Stopped: No beneficial effects on biomarker or clinical efficacy endpoints in the VGL101-01.201 Study
Sponsor: Vigil Neuroscience, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: VGL101-01.002
Record Dates: First submitted 2021-08-18; First posted 2021-08-25 (Actual); Results first posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-07

CONDITIONS: ALSP
Keywords: ALSP; CSF1R; leukoencephalopathy; Hereditary Diffuse Leukoencephalopathy with Spheroids; HDLS; CSF1R-related Leukoencephalopathy; Adult-Onset Leukoencephalopathy with Axonal Spheroids and Pigmented Glia; CSF1R gene mutation; POLD; Pigmentary Orthochromatic Leukodystrophy
MeSH Terms: conditions — Leukoencephalopathies; Hereditary Diffuse Leukoencephalopathy with Spheroids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with ALSP
  Interventions: Other: No intervention
- Patients with Prodromal ALSP
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Not applicable for a Natural History Study

SUMMARY:
Adult-onset leukoencephalopathy with axonal spheroids and pigmented glia (ALSP) is a rare, rapidly progressing, genetic, neurodegenerative disease for which no definitive treatment options and limited information on the natural history of the disease are available. The structural, genetic, and neuropathophysiological abnormalities of ALSP lead to the onset of neurologic symptoms, such as moderate to severe motor and neuropsychiatric impairments. This natural history study will collect data to contribute to the development of future novel therapies that focus on the neuropathophysiological features that underlie ALSP and that are essential to reverse, delay, or stop progression of this debilitating disorder.

ELIGIBILITY:
Key Inclusion Criteria for Definitive ALSP patients:

1. Subjects who have documentation of a gene mutation in the CSF1R gene (prior to enrollment)
2. Subjects who fulfill both of the following criteria (a and b):

   a. More than two findings of clinical signs or symptoms in the following categories: i. Cognitive impairment or psychiatric problem ii. Pyramidal signs on neurological examination iii. Extrapyramidal signs, such as rigidity, tremor, abnormal gait, or bradykinesia iv. Epilepsy

   b. MRI findings consistent with ALSP: specifically, bilateral cerebral white matter lesions with or without thinning of the corpus callosum NOTE: Subjects with other causes of leukoencephalopathy, including vascular dementia, multiple sclerosis, or leukodystrophy (e.g., adrenoleukodystrophy, Krabbe disease, metachromatic leukodystrophy), will be excluded.
3. Subjects who, in the investigator's opinion, have demonstrated clinical progression of their ALSP within the past year.
4. Subjects who meet the criteria for definitive ALSP must have a designated study partner (i.e caregiver) who spends at least 4 hours per week with them. The study partner must be able and willing to assist the subject in complying with the study requirements, be able to provide information during study visits, and be willing to sign a study partner ICF. Subjects who do not have a study partner may be enrolled at the investigator's discretion if they are able to comply with protocol requirements.

Key Exclusion Criteria for Definitive ALSP patients:

1. Subjects with any neurological or psychiatric diseases that can produce cognitive, motor, or behavioral impairment similar to ALSP, including, but not limited to, Alzheimer's disease, frontotemporal dementia, ALS, stroke, Huntington disease, multiple sclerosis, Parkinson's disease, and Down syndrome, or with active alcohol/drug abuse
2. Subjects who are unable to undergo MRI
3. Subjects with any condition or situation that, in the opinion of the investigator or sponsor medical personnel, may place the subject at significant risk, confound the study results, or interfere significantly with the subject's participation in the study.
4. Subjects who have previously undergone HSCT or plan to undergo HSCT within 12 months of the Screening/Baseline visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Definitive ALSP and Prodromal ALSP.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (6):
  - Investigative Site 4, San Francisco, California
  - Investigative Site 5, Englewood, Colorado
  - Investigative Site 1, Boca Raton, Florida
  - Investigative Site 2, Jacksonville, Florida
  - Investigative Site 11, Boston, Massachusetts
  - Investigative Site 10, Philadelphia, Pennsylvania
- Investigative Site 12, São Paulo, Brazil
- Investigative Site 3, London, Ontario, Canada
- Germany (2):
  - Investigative Site 8, Leipzig
  - Investigative Site 9, Tübingen
- Investigative Site 6, Amsterdam, Netherlands
- Investigative Site 7, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 11 sites that screened participants in the United States, Canada, Netherlands, United Kingdom, Germany, and Brazil. The first participant was enrolled on September 13, 2021 and the last participant was enrolled on April 23, 2025.
Pre-assignment Details: Of 82 screened patients, 26 failed to meet eligibility criteria. Of 56 participants enrolled in the study, 53 were enrolled prior to the data cutoff of February 19, 2025.
Groups:
- Prodromal: ALSP participants with confirmed CSF1R mutation, radiographic evidence of ALSP, and who had none or up to and including 2 ALSP-related clinical signs or symptoms.
- Symptomatic/Definitive ALSP (no HSCT): ALSP participants with confirmed CSF1R mutation, radiographic evidence of ALSP and had at least 3 ALSP-related clinical signs or symptoms, and did not have hematopoietic stem cell transplant (HSCT) procedure.
- Symptomatic/Definitive ALSP (Prior HSCT): ALSP participants with CSF1R mutation, radiographic evidence of ALSP and had at least 3 ALSP-related clinical signs or symptoms, and had prior hematopoietic stem cell transplant (HSCT) procedure.
Period: Overall Study
Arm/Group | Prodromal | Symptomatic/Definitive ALSP (no HSCT) | Symptomatic/Definitive ALSP (Prior HSCT)
Started | 19 | 23 | 11
Completed | 6 | 0 | 0
Not Completed | 13 | 23 | 11
Not completed — Enrollment in Interventional Study | 2 | 9 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Study Termination by Sponsor | 10 | 11 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prodromal | Symptomatic/Definitive ALSP (no HSCT) | Symptomatic/Definitive ALSP (Prior HSCT) | Total
Number analyzed (Participants) | 19 | 23 | 11 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (16.62) | 44.5 (11.54) | 47.5 (4.55) | 45.4 (12.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 4 | 31
  Male | 7 | 8 | 7 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 0 | 4
  White | 18 | 19 | 10 | 47
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 6 | 1 | 9
  Not Hispanic or Latino | 17 | 16 | 10 | 43
  Unknown or Not Reported | 0 | 1 | 0 | 1
Age at Diagnosis [Mean (Standard Deviation); unit: years] — Age of participant when ALSP was diagnosed Population: 9 prodromal and 1 symptomatic/definitive ALSP (no HSCT) subjects had unknown age of diagnosis.
  years
    number analyzed (Participants) | 10 | 22 | 11 | 43
    (all) | 45.0 (15.00) | 43.6 (11.18) | 43.9 (4.60) | 44.0 (10.78)
Duration Since Diagnosis [Mean (Standard Deviation); unit: years] — Duration of time from ALSP diagnosis to study entry Population: 9 prodromal and 1 symptomatic/definitive ALSP (no HSCT) subjects had unknown age of diagnosis.
  years
    number analyzed (Participants) | 10 | 22 | 11 | 43
    (all) | 1.1 (1.29) | 1.0 (1.40) | 4.1 (1.46) | 1.8 (1.92)

OUTCOME MEASURES:

1. Primary Outcome: Magnetic Resonance Imaging (MRI) Ventricle Volume
Description: Change from Baseline in ventricle volume at Month 6
Time Frame: Month 6
Population: Not all participants completed Month 6 visit prior to data cutoff.
Measure: Mean (Standard Deviation); unit: cubic millimeter
Arm/Group | Prodromal | Symptomatic/Definitive ALSP (no HSCT) | Symptomatic/Definitive ALSP (Prior HSCT)
Number analyzed (Participants) | 18 | 14 | 10
cubic millimeter | 498.3 (833.03) | 4153.2 (6052.35) | 3061.5 (5142.76)

2. Primary Outcome: Magnetic Resonance Imaging (MRI) Ventricle Volume
Description: Change from Baseline in ventricle volume at Month 12
Time Frame: Month 12
Population: Not all participants completed Month 12 visit prior to data cutoff.
Measure: Mean (Standard Deviation); unit: cubic millimeter
Arm/Group | Prodromal | Symptomatic/Definitive ALSP (no HSCT) | Symptomatic/Definitive ALSP (Prior HSCT)
Number analyzed (Participants) | 18 | 7 | 9
cubic millimeter | 1030.5 (1409.76) | 10410.0 (7798.42) | 3565.6 (8930.46)

3. Primary Outcome: Magnetic Resonance Imaging (MRI) Ventricle Volume
Description: Change from Baseline in ventricle volume at Month 18
Time Frame: Month 18
Population: Not all participants completed Month 18 visit prior to data cutoff.
Measure: Mean (Standard Deviation); unit: cubic millimeter
Arm/Group | Prodromal | Symptomatic/Definitive ALSP (no HSCT) | Symptomatic/Definitive ALSP (Prior HSCT)
Number analyzed (Participants) | 17 | 2 | 8
cubic millimeter | 1236.9 (2139.02) | 17758.8 (17376.19) | 5462.0 (6719.45)

4. Primary Outcome: Magnetic Resonance Imaging (MRI) Ventricle Volume
Description: Change from Baseline in ventricle volume at Month 24
Time Frame: Month 24
Population: Not all participants completed Month 24 visit prior to data cutoff.
Measure: Mean (Standard Deviation); unit: cubic millimeter
Arm/Group | Prodromal | Symptomatic/Definitive ALSP (no HSCT) | Symptomatic/Definitive ALSP (Prior HSCT)
Number analyzed (Participants) | 11 | 1 | 9
cubic millimeter | 1216.8 (2013.70) | 8901.6 (NA) — only 1 value | 5406.7 (5977.76)

5. Primary Outcome: Magnetic Resonance Imaging (MRI) Ventricle Volume
Description: Change from Baseline in ventricle volume at Month 30
Time Frame: Month 30
Population: Not all participants completed Month 30 visit prior to data cutoff.
Measure: Mean (Standard Deviation); unit: cubic millimeter
Arm/Group | Prodromal | Symptomatic/Definitive ALSP (no HSCT) | Symptomatic/Definitive ALSP (Prior HSCT)
Number analyzed (Participants) | 6 | 1 | 4
cubic millimeter | 1837.6 (2931.17) | 13821.3 (NA) — only 1 value | 9115.2 (8421.27)

ADVERSE EVENTS:
Time Frame: From the time of signing the informed consent through up to 36 months
Description: For this observational study, an adverse event was defind as any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may not be considered related to a study procedure.
Arm/Group | Prodromal | Symptomatic/Definitive ALSP (no HSCT) | Symptomatic/Definitive ALSP (Prior HSCT)
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/23 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/19 | 2/23 | 1/11
Other Adverse Events (participants affected / at risk) | 7/19 | 6/23 | 4/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prodromal (N=19) | Symptomatic/Definitive ALSP (no HSCT) (N=23) | Symptomatic/Definitive ALSP (Prior HSCT) (N=11)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prodromal (N=19) | Symptomatic/Definitive ALSP (no HSCT) (N=23) | Symptomatic/Definitive ALSP (Prior HSCT) (N=11)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Contrast media allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (4) | 0 (0)
Facial asymmetry (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Migraine without aura (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Uriinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-10-02): https://cdn.clinicaltrials.gov/large-docs/43/NCT05020743/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-19): https://cdn.clinicaltrials.gov/large-docs/43/NCT05020743/SAP_001.pdf